CLINICAL TRIAL: NCT05464420
Title: A Phase 3 Randomized, Double-blind, Active Comparator-controlled, Lot-to-Lot Consistency Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Adults 18 to 49 Years of Age
Brief Title: A Study to Evaluate the Safety, Tolerability, Immunogenicity, and Lot Consistency of V116 in Adults 18 to 49 Years of Age (V116-004, STRIDE-4)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V116-004; 2022-000265-41 (EudraCT Number)
Record Dates: First submitted 2022-07-12; First posted 2022-07-19 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- V116 Lot 1 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) dose of V116 Lot 1 on Day 1.
  Interventions: Biological: V116
- V116 Lot 2 (Experimental): Participants will receive a single 0.5 mL IM dose of V116 Lot 2 on Day 1.
  Interventions: Biological: V116
- V116 Lot 3 (Experimental): Participants will receive a single 0.5 mL IM dose of V116 Lot 3 on Day 1.
  Interventions: Biological: V116
- PPSV23 (Active Comparator): Participants will receive a single 0.5 mL IM dose of PPSV23 on Day 1.
  Interventions: Biological: PPSV23

INTERVENTIONS:
Biological: V116 — Pneumococcal 21-valent conjugate vaccine with 4 μg of each of the following pneumococcal polysaccharides (PnPs) antigen: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B in each 0.5 mL sterile solution
  Other Names: Pneumococcal 21-valent Conjugate Vaccine
  Arms: V116 Lot 1; V116 Lot 2; V116 Lot 3
Biological: PPSV23 — Pneumococcal 23-valent conjugate vaccine with 25 μg of each of the following PnPs antigen: 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in each 0.5 mL sterile solution
  Other Names: PNEUMOVAX™23
  Arms: PPSV23

SUMMARY:
This study will evaluate the safety, tolerability, and immunogenicity of a pneumococcal 21-valent conjugate vaccine (V116) in pneumococcal vaccine-naïve adults 18 to 49 years of age.

The primary study hypothesis is that all 3 lots of V116 are equivalent as assessed by the serotype-specific opsonophagocytic activity (OPA) Geometric Mean Titers (GMTs) at 30 days postvaccination for all serotypes included in V116.

ELIGIBILITY:
The key inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has underlying chronic conditions but assessed to be stable as per investigator
* Has ability to complete electronic Vaccine Report Card (eVRC) data collection without assistance as per investigator

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (IPD) or other culture-positive pneumococcal disease ≤3 years before Visit 1 (Day 1)
* Has a known or suspected congenital immunodeficiency, functional or anatomic asplenia, or history of autoimmune disease
* Has a coagulation disorder contraindicating intramuscular vaccination
* Has a recent illness with fever
* Has a known malignancy that is progressing or has required active treatment <3 years before enrollment
* Is expected to receive any pneumococcal vaccine during the study outside of the protocol
* Has received systemic corticosteroids for ≥14 consecutive days and has not completed treatment ≥14 days before receipt of study vaccine
* Is currently receiving immunosuppressive therapy, including chemotherapeutic agents or other immunotherapies/immunomodulators used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Has received any non-live vaccine ≤14 days before receipt of study vaccine or is scheduled to receive any non-live vaccine ≤30 days after receipt of study vaccine
* Has received any live vaccine ≤30 days before receipt of study vaccine or is scheduled to receive any live vaccine ≤30 days after receipt of study vaccine
* Has received a blood transfusion or blood products, including immunoglobulins ≤6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product ≤30 days after receipt of study vaccine

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2162 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (72):
- United States (30):
  - Desert Clinical Research/ CCT Research ( Site 0019), Mesa, Arizona
  - Fiel Family and Sports Medicine, PC/CCT Research ( Site 0008), Tempe, Arizona
  - Baptist Health Center For Clinical Research ( Site 0015), Little Rock, Arkansas
  - Valley Clinical Trials, Inc. ( Site 0023), Northridge, California
  - Artemis Institute for Clinical Research ( Site 0027), San Diego, California
  - Millennium Clinical Trials ( Site 0004), Simi Valley, California
  - Diablo Clinical Research, Inc. ( Site 0022), Walnut Creek, California
  - Lynn Institute of Denver ( Site 0003), Aurora, Colorado
  - Indago Research & Health Center, Inc ( Site 0011), Hialeah, Florida
  - L&C Professional Medical Research Institute ( Site 0012), Miami, Florida
  - Headlands Research Orlando ( Site 0017), Orlando, Florida
  - Clinical Research Trials of Florida ( Site 0001), Tampa, Florida
  - Clinical Research Prime Rexburg ( Site 0040), Rexburg, Idaho
  - Healthcare Research Network - Chicago ( Site 0006), Flossmoor, Illinois
  - Kentucky Pediatric/ Adult Research ( Site 0036), Bardstown, Kentucky
  - Alliance for Multispecialty Research, LLC ( Site 0031), Kansas City, Missouri
  - Methodist Physicians Clinic/CCT Research ( Site 0029), Fremont, Nebraska
  - Healor Primary Care / CCT Research ( Site 0028), Las Vegas, Nevada
  - Axces Research ( Site 0034), Santa Fe, New Mexico
  - Rochester Clinical Research, Inc. ( Site 0033), Rochester, New York
  - M3 Wake Research Associates ( Site 0035), Raleigh, North Carolina
  - Lynn Health Science Institute ( Site 0014), Oklahoma City, Oklahoma
  - Velocity Clinical Research, Providence ( Site 0018), East Greenwich, Rhode Island
  - Velocity Clinical Research, Greenville ( Site 0021), Greenville, South Carolina
  - Clinical Research Associates Inc ( Site 0039), Nashville, Tennessee
  - DCOL Center for Clinical Research ( Site 0025), Longview, Texas
  - IMA Clinical Research San Antonio ( Site 0020), San Antonio, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research ( Site 0016), Tomball, Texas
  - Charlottesville Medical Research ( Site 0013), Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc. ( Site 0002), Newport News, Virginia
- Austria (4):
  - Medizinische Universität Graz-Klinische Abteilung für Pulmonologie ( Site 0304), Graz, Styria
  - Medizinische Universitaet Innsbruck ( Site 0301), Innsbruck, Tyrol
  - Tropeninstitut Wien 1060 ( Site 0300), Vienna, Vienna
  - Medizinische Universität Wien ( Site 0302), Vienna
- Canada (8):
  - Colchester Research Group ( Site 0202), Truro, Nova Scotia
  - Hamilton Medical Research Group ( Site 0208), Hamilton, Ontario
  - Milestone Research Inc. ( Site 0201), London, Ontario
  - Manna Research Toronto ( Site 0209), Toronto, Ontario
  - Manna Research Mirabel ( Site 0207), Mirabel, Quebec
  - Manna Research Montreal ( Site 0203), Pointe-Claire, Quebec
  - Q&T Research Sherbrooke Inc. ( Site 0204), Sherbrooke, Quebec
  - Diex Recherche Trois-Rivieres ( Site 0206), Trois-Rivières, Quebec
- Denmark (5):
  - Sanos Clinic-Sanos Clinic ( Site 0402), Herlev, Capital Region
  - Danske Lægers Vaccinations Service - Søborg ( Site 0404), Søborg, Capital Region
  - Danske Lægers Vaccinations Service - Århus ( Site 0403), Aarhus, Central Jutland
  - Sanos Clinic - Nordjylland ( Site 0401), Aalborg, North Denmark
  - Sanos Clinic - Syddanmark ( Site 0400), Vejle, Region Syddanmark
- Finland (7):
  - FVR, Oulun rokotetutkimusklinikka ( Site 0501), Oulu, North Ostrobothnia
  - FVR, Porin rokotetutkimusklinikka ( Site 0508), Pori, Satakunta
  - FVR, Seinäjoen rokotetutkimusklinikka ( Site 0504), Seinäjoki, South Ostrobothnia
  - FVR, Turun rokotetutkimusklinikka ( Site 0500), Turku, Southwest Finland
  - FVR, Espoon rokotetutkimusklinikka ( Site 0509), Espoo, Uusimaa
  - FVR, Etelä-Helsingin rokotetutkimusklinikka ( Site 0503), Helsinki, Uusimaa
  - Helsinki East Vaccine Research Clinic ( Site 0502), Helsinki, Uusimaa
- Israel (6):
  - Rambam Health Care Campus ( Site 0603), Haifa
  - Maccabi Healthcare Services ( Site 0606), Jerusalem
  - Hadassah Medical Center ( Site 0600), Jerusalem
  - Meir Medical Center ( Site 0601), Kfar Saba
  - Sheba Medical Center-Early Phase Clinical Trials Unit ( Site 0604), Ramat Gan
  - Clalit Health Services - Sakhnin Community Clinic-Research Unit ( Site 0602), Sakhnin
- Poland (6):
  - IN VIVO ( Site 0711), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Pratia Bydgoszcz-Centrum Medyczne Pratia Bydgoszcz ( Site 0709), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun ( Site 0706), Torun, Kuyavian-Pomeranian Voivodeship
  - Alergotest s.c Specjalistyczne Centrum Medyczne ( Site 0703), Lublin, Lublin Voivodeship
  - Centrum Medyczne Medyk ( Site 0704), Rzeszów, Podkarpackie Voivodeship
  - Clinmedica OMC ( Site 0701), Skierniewice, Łódź Voivodeship
- Spain (6):
  - EBA CENTELLES ( Site 0800), Centelles, Catalonia
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-Respiratory ( Site 0808), Pozuelo de Alarcón, Madrid
  - Fundación Oftalmologica del Mediterraneo-Vaccine Research ( Site 0818), Valencia, Valenciana, Comunitat
  - Centre d'Atenció Primària Vallcarca - Sant Gervasi ( Site 0801), Barcelona
  - EAP Sardenya ( Site 0802), Barcelona
  - Hospital La Princesa-Clinical Pharmacology ( Site 0815), Madrid

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Scott P, Ukkonen B, Caraco Y, Perez SN, Alpizar SA, Cardona JF, Greenberg D, Grijalva CG, Orenstein W, Wiedmann RT, Fernsler D, Cheon K, Li J, Platt HL. A phase 3, randomized trial to evaluate lot-to-lot consistency of V116, an adult-specific pneumococcal conjugate vaccine (STRIDE-4). Med. 2025 Oct 10;6(10):100748. doi: 10.1016/j.medj.2025.100748. Epub 2025 Jun 20. PMID 40543503
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26086&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy pneumococcal vaccine-naïve adults between 18 and 49 years of age were enrolled in this study.
Groups:
- V116 Lot 1: Participants received a single 0.5 mL intramuscular (IM) dose of V116 Lot 1 on Day 1.
- V116 Lot 2: Participants received a single 0.5 mL IM dose of V116 Lot 2 on Day 1.
- V116 Lot 3: Participants received a single 0.5 mL IM dose of V116 Lot 3 on Day 1.
- PPSV23: Participants received a single 0.5 mL IM dose of PPSV23 on Day 1.
Period: Overall Study
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Started | 541 | 540 | 541 | 540
Vaccinated | 539 | 538 | 540 | 540
Safety Analysis Population (One participant initially randomized to the V116 Lot 2 arm received V116 Lot 1, one participant initially randomized to the V116 Lot 1 arm received V116 Lot 3, and one participant initially randomized to the V116 Lot 2 arm received PPSV23.) | 539 | 536 | 541 | 541
Completed | 521 | 520 | 525 | 526
Not Completed | 20 | 20 | 16 | 14
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 16 | 11 | 11 | 11
Not completed — Randomized in Error Without Study Treatment | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 3 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Unable to Adhere to Study Schedule | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23 | Total
Number analyzed (Participants) | 541 | 540 | 541 | 540 | 2162
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (9.3) | 34.8 (9.2) | 34.3 (9.3) | 34.4 (9.2) | 34.6 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305 | 321 | 311 | 310 | 1247
  Male | 236 | 219 | 230 | 230 | 915
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 98 | 104 | 113 | 107 | 422
  Not Hispanic or Latino | 440 | 434 | 420 | 430 | 1724
  Unknown or Not Reported | 3 | 2 | 8 | 3 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 2 | 4 | 4 | 16
  Asian | 9 | 12 | 6 | 8 | 35
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 1 | 4
  Black or African American | 49 | 43 | 55 | 48 | 195
  White | 458 | 458 | 458 | 453 | 1827
  More than one race | 16 | 24 | 16 | 26 | 82
  Unknown or Not Reported | 1 | 0 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-site Adverse Events (AEs) Following Vaccination With Separate V116 Lots
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs included pain/tenderness, redness/erythema, and swelling. Per protocol, the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Up to 5 days
Population: Per protocol, all randomized participants who received one of three lots of V116 were analyzed according to the vaccination they received. One participant randomized to the V116 Lot 1 incorrectly received V116 Lot 3 and one participant randomized into the V116 Lot 2 group incorrectly received V116 Lot 1, and one participant randomized to the V116 Lot 2 arm incorrectly received PPSV23.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 536 | 541 | 0
Percentage of Participants
  Injection site erythema | 13.4 [10.6 to 16.5] | 14.2 [11.3 to 17.4] | 13.1 [10.4 to 16.3] |
  Injection site pain | 72.9 [68.9 to 76.6] | 72.9 [69.0 to 76.7] | 73.9 [70.0 to 77.6] |
  Injection site swelling | 12.4 [9.8 to 15.5] | 15.3 [12.4 to 18.6] | 11.8 [9.2 to 14.9] |

2. Primary Outcome: Percentage of Participants With Solicited Injection-site AEs Following Vaccination: Combined Lots of V116 or PPSV23
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection-site AEs included pain/tenderness, redness/erythema, and swelling. Per the statistical analysis plan, no within group method of dispersion (MOD) were planned or calculated.
Time Frame: Up to 5 days
Population: All randomized participants who received study vaccination were analyzed according to the vaccination they received. One participant randomized into the V116 Lot 2 group incorrectly received PPSV23.
Measure: Number; unit: Percentage of Participants
Groups:
- V116 Combined Lots 1, 2, and 3: Participants received a single 0.5 mL IM dose of either V116 Lot 1, 2, or 3 on Day 1.
Arm/Group | V116 Combined Lots 1, 2, and 3 | PPSV23
Number analyzed (Participants) | 1616 | 541
Percentage of Participants
  Injection site erythema | 13.6 | 7.6
  Injection site pain | 73.3 | 60.6
  Injection site swelling | 13.2 | 7.6
Statistical Analysis 1: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Injection site erythema: V116 Combined Lots - PPSV23; Test type: Other — Estimated difference in percentage and 95% confidence intervals (CI) were based on the Miettinen & Nurminen method; Estimated difference in percentage = 6.0, 95% CI 2-sided [3.0 to 8.6]
Statistical Analysis 2: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Injection site pain: V116 Combined Lots - PPSV23; Test type: Other — Estimated difference in percentage and 95% CI were based on the Miettinen & Nurminen method; Estimated difference in percentage = 12.6, 95% CI 2-sided [8.0 to 17.3]
Statistical Analysis 3: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Injection site swelling: V116 Combined Lots - PPSV23; Test type: Other — Estimated difference in percentage and 95% CI were based on the Miettinen & Nurminen method; Estimated difference in percentage = 5.6, 95% CI 2-sided [2.6 to 8.2]

3. Primary Outcome: Percentage of Participants With Solicited Systemic AEs Following Vaccination With Separate V116 Lots
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs included headache, muscle aches/myalgia, tiredness/fatigue, and pyrexia. Per protocol, the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Up to 5 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 536 | 541 | 0
Percentage of Participants
  Fatigue | 38.0 [33.9 to 42.3] | 34.0 [30.0 to 38.1] | 34.4 [30.4 to 38.6] |
  Headache | 28.0 [24.3 to 32.0] | 26.1 [22.4 to 30.1] | 27.5 [23.8 to 31.5] |
  Myalgia | 18.2 [15.0 to 21.7] | 13.6 [10.8 to 16.8] | 17.2 [14.1 to 20.6] |
  Pyrexia | 3.2 [1.8 to 5.0] | 2.2 [1.2 to 3.9] | 3.5 [2.1 to 5.4] |

4. Primary Outcome: Percentage of Participants With Solicited Systemic AEs Following Vaccination: Combined Lots of V116 or PPSV23
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs included headache, muscle aches/myalgia, tiredness/fatigue, and pyrexia. Per the statistical analysis plan, no within group method of dispersion (MOD) were planned or calculated.
Time Frame: Up to 5 days
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | V116 Combined Lots 1, 2, and 3 | PPSV23
Number analyzed (Participants) | 1616 | 541
Percentage of Participants
  Fatigue | 35.5 | 34.0
  Headache | 27.2 | 21.4
  Myalgia | 16.3 | 8.7
  Pyrexia | 3.0 | 2.2
Statistical Analysis 1: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Fatigue: V116 Combined Lots - PPSV23; Test type: Other — Estimated difference in percentage and 95% CI were based on the Miettinen & Nurminen method; Estimated difference in percentage = 1.4, 95% CI 2-sided [-3.2 to 6.0]
Statistical Analysis 2: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Headache: V116 Combined Lots - PPSV23; Test type: Other — Estimated difference in percentage and 95% CI were based on the Miettinen & Nurminen method; Estimated difference in percentage = 5.8, 95% CI 2-sided [1.6 to 9.7]
Statistical Analysis 3: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Myalgia: V116 Combined Lots - PPSV23; Test type: Other — Estimated difference in percentage and 95% CI were based on the Miettinen & Nurminen method; Estimated difference in percentage = 7.6, 95% CI 2-sided [4.5 to 10.5]
Statistical Analysis 4: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Pyrexia: V116 Combined Lots - PPSV23; Test type: Other — Estimated difference in percentage and 95% CI were based on the Miettinen & Nurminen method; Estimated difference in percentage = 0.8, 95% CI 2-sided [-1.0 to 2.1]

5. Primary Outcome: Percentage of Participants With Vaccine-related Serious Adverse Events (SAEs) Following Vaccination With Separate V116 Lots
Description: An SAE was any untoward medical occurrence that, at any dose, resulted in death, was life threatening, required inpatient hospitalization or prolonged existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was another important medical event. SAEs that were reported to be at least possibly related by the investigator to study vaccination were reported. Per protocol, the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Up to 194 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 536 | 541 | 0
Percentage of Participants | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.7] | 0.0 [0.0 to 0.7] |

6. Primary Outcome: Percentage of Participants With Vaccine-related SAEs Following Vaccination: Combined Lots of V116 or PPSV23
Description: An SAE was any untoward medical occurrence that, at any dose, resulted in death, was life threatening, required inpatient hospitalization or prolonged existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was another important medical event. SAEs that were reported to be at least possibly related by the investigator to study vaccination were reported. Per the statistical analysis plan, no within group MOD were planned or calculated.
Time Frame: Up to 194 days
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | V116 Combined Lots 1, 2, and 3 | PPSV23
Number analyzed (Participants) | 1616 | 541
Percentage of Participants | 0.0 | 0.0
Statistical Analysis 1: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Vaccine-related SAEs: V116 Combined Lots - PPSV23; Test type: Other — Estimated difference in percentage and 95% CI were based on the Miettinen & Nurminen method; Estimated difference in percentage = 0.0, 95% CI 2-sided [-0.7 to 0.2]

7. Primary Outcome: Geometric Mean Titers (GMTs) of Serotype-specific Opsonophagocytic Activity (OPA) for All Serotypes in V116 Following Vaccination With Separate V116 Lots
Description: Serotype-specific OPA titers for all serotypes in V116 following vaccination were determined using multiplex opsonophagocytic assay (MOPA). Serotype-specific OPA GMTs and GMT ratios with 95% confidence intervals (CIs) were calculated using a constrained longitudinal data analysis (cLDA) model. Per protocol, within-group CIs were not calculated and the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Day 30
Population: Per protocol, all randomized participants who were vaccinated with V116 and were without deviations from the protocol that may substantially affect the results of the immunogenicity endpoint and who had sufficient data to perform the analysis. Deviations include, but are not limited to the following: randomized but not vaccinated, blood drawn out of time window, prohibited concomitant medication or vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 538 | 540 | 0
Titers
  Serotype 3: number analyzed (Participants) | 524 | 525 | 525 | 0
  Serotype 3 | 327.2 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 299.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 318.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 6A: number analyzed (Participants) | 515 | 523 | 524 | 0
  Serotype 6A | 6901.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6014.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6641.2 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 7F: number analyzed (Participants) | 522 | 531 | 527 | 0
  Serotype 7F | 7219.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6201.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6657.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 8: number analyzed (Participants) | 527 | 530 | 528 | 0
  Serotype 8 | 3935.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3812.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3765.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 9N: number analyzed (Participants) | 526 | 533 | 531 | 0
  Serotype 9N | 18747.4 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 17201.6 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 18557.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 10A: number analyzed (Participants) | 524 | 529 | 533 | 0
  Serotype 10A | 7570.2 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7796.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7330.4 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 11A: number analyzed (Participants) | 518 | 531 | 532 | 0
  Serotype 11A | 6396.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6630.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6374.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 12F: number analyzed (Participants) | 523 | 532 | 528 | 0
  Serotype 12F | 7478.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6803.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7329.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 15A: number analyzed (Participants) | 502 | 505 | 513 | 0
  Serotype 15A | 10698.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10253.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10692.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 15C: number analyzed (Participants) | 522 | 527 | 522 | 0
  Serotype 15C | 13133.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11441.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11177.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 16F: number analyzed (Participants) | 521 | 521 | 521 | 0
  Serotype 16F | 9239.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9550.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9530.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 17F: number analyzed (Participants) | 525 | 531 | 532 | 0
  Serotype 17F | 17185.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 17718.6 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 16886.7 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 19A: number analyzed (Participants) | 527 | 533 | 533 | 0
  Serotype 19A | 3187.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3123.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3368.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 20A: number analyzed (Participants) | 524 | 525 | 525 | 0
  Serotype 20A | 16339.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 16676.2 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 15302.4 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 22F: number analyzed (Participants) | 521 | 523 | 529 | 0
  Serotype 22F | 11638.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10614.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11346.7 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 23A: number analyzed (Participants) | 509 | 521 | 520 | 0
  Serotype 23A | 8437.4 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8459.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8322.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 23B: number analyzed (Participants) | 526 | 530 | 527 | 0
  Serotype 23B | 2964.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2435.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3035.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 24F: number analyzed (Participants) | 522 | 522 | 524 | 0
  Serotype 24F | 4861.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4783.4 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4758.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 31: number analyzed (Participants) | 516 | 527 | 522 | 0
  Serotype 31 | 9052.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8831.6 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8870.7 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 33F: number analyzed (Participants) | 521 | 529 | 526 | 0
  Serotype 33F | 37994.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 34227.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 35182.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 35B: number analyzed (Participants) | 523 | 528 | 527 | 0
  Serotype 35B | 12971.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 12586.6 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 12494.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
Statistical Analysis 1: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 3: GMT Ratio V116 Lot 1/ V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; P value for testing the lower bound of the 95% CI for GMT ratio was >0.5. P value for testing the upper bound of the 95% CI for GMT ratio was <2.0; GMT Ratio = 1.09, 95% CI 2-sided [0.96 to 1.24] — V116 Lot 1/V116 Lot 2
Statistical Analysis 2: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 3: GMT Ratio V116 Lot 1/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.03, 95% CI 2-sided [0.90 to 1.17] — V116 Lot 1/ V116 Lot 3
Statistical Analysis 3: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 3: GMT Ratio V116 Lot 2/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA Model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.94, 95% CI 2-sided [0.83 to 1.06] — V116 Lot 2/ V116 Lot 3
Statistical Analysis 4: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 6A: GMT Ratio V116 Lot 1/ V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.15, 95% CI 2-sided [0.97 to 1.35] — V116 Lot 1/V116 Lot 2
Statistical Analysis 5: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 6A: GMT Ratio V116 Lot 1/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.04, 95% CI 2-sided [0.88 to 1.22] — V116 Lot 1/V116 Lot 3
Statistical Analysis 6: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 6A: GMT Ratio V116 Lot 2/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.91, 95% CI 2-sided [0.77 to 1.06] — V116 Lot 2/V116 Lot 3
Statistical Analysis 7: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 7F: V116 Lot 1/ V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.16, 95% CI 2-sided [1.01 to 1.34] — V116 Lot 1/V116 Lot 2
Statistical Analysis 8: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 7F: GMT Ratio V116 Lot 1/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.08, 95% CI 2-sided [0.94 to 1.25] — V116 Lot 1/V116 Lot 3
Statistical Analysis 9: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 7F: GMT Ratio V116 Lot 2/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.93, 95% CI 2-sided [0.81 to 1.07] — V116 Lot 2/V116 Lot 3
Statistical Analysis 10: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 8 V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.03, 95% CI 2-sided [0.92 to 1.16] — V116 Lot 1/V116 Lot 2
Statistical Analysis 11: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 8: GMT Ratio V116 Lot 1/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.05, 95% CI 2-sided [0.93 to 1.18] — V116 Lot 1/ V116 Lot 3
Statistical Analysis 12: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 8: GMT Ratio V116 Lot 2/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.01, 95% CI 2-sided [0.90 to 1.14] — V116 Lot 2/ V116 Lot 3
Statistical Analysis 13: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 9N: GMT Ratio V116 Lot 1/ V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.09, 95% CI 2-sided [0.94 to 1.26] — V116 Lot 1/V116 Lot 2
Statistical Analysis 14: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 9N: GMT Ratio V116 Lot 1/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.01, 95% CI 2-sided [0.87 to 1.17] — V116 Lot 1/V116 Lot 3
Statistical Analysis 15: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 9N: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.93, 95% CI 2-sided [0.80 to 1.07] — V116 Lot 2/V116 Lot 3
Statistical Analysis 16: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 10A: GMT Ratio V116 Lot 1/ V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.97, 95% CI 2-sided [0.85 to 1.11] — V116 Lot 1/V116 Lot 2
Statistical Analysis 17: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 10A: GMT Ratio V116 Lot 1/ V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.03, 95% CI 2-sided [0.91 to 1.18] — V116 Lot 1/V116 Lot 3
Statistical Analysis 18: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 10A: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.06, 95% CI 2-sided [0.93 to 1.21] — V116 Lot 2/V116 Lot 3
Statistical Analysis 19: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 11A: GMT Ratio V116 Lot 1/ V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.96, 95% CI 2-sided [0.84 to 1.11] — V116 Lot 1/V116 Lot 2
Statistical Analysis 20: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 11A: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.87 to 1.16] — V116 Lot 1/V116 Lot 3
Statistical Analysis 21: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 11A: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.04, 95% CI 2-sided [0.90 to 1.20] — V116 Lot 2/V116 Lot 3
Statistical Analysis 22: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 12F: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.10, 95% CI 2-sided [0.96 to 1.26] — V116 Lot 1/V116 Lot 2
Statistical Analysis 23: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 12F: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.89 to 1.17] — V116 Lot 1/V116 Lot 3
Statistical Analysis 24: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 12F: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.93, 95% CI 2-sided [0.81 to 1.07] — V116 Lot 2/V116 Lot 3
Statistical Analysis 25: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 15A: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.04, 95% CI 2-sided [0.89 to 1.22] — V116 Lot 1/V116 Lot 2
Statistical Analysis 26: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 15A: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.86 to 1.17] — V116 Lot 1/V116 Lot 3
Statistical Analysis 27: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 15A: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.96, 95% CI 2-sided [0.82 to 1.12] — V116 Lot 2/V116 Lot 3
Statistical Analysis 28: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 15C: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.15, 95% CI 2-sided [0.95 to 1.38] — V116 Lot 1/V116 Lot 2
Statistical Analysis 29: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 15C: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.18, 95% CI 2-sided [0.97 to 1.42] — V116 Lot 1/V116 Lot 3
Statistical Analysis 30: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 15C: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.85 to 1.23] — V116 Lot 2/V116 Lot 3
Statistical Analysis 31: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 16F: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.97, 95% CI 2-sided [0.84 to 1.11] — V116 Lot 1/V116 Lot 2
Statistical Analysis 32: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 16F: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.97, 95% CI 2-sided [0.84 to 1.11] — V116 Lot 1/V116 Lot 3
Statistical Analysis 33: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 16F: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.87 to 1.15] — V116 Lot 2/V116 Lot 3
Statistical Analysis 34: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 17F: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.97, 95% CI 2-sided [0.85 to 1.11] — V116 Lot 1/V116 Lot 2
Statistical Analysis 35: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 17F: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.89 to 1.17] — V116 Lot 1/V116 Lot 3
Statistical Analysis 36: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 17F: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.05, 95% CI 2-sided [0.92 to 1.20] — V116 Lot 2/V116 Lot 3
Statistical Analysis 37: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 19A: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.91 to 1.15] — V116 Lot 1/V116 Lot 2
Statistical Analysis 38: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 19A: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.95, 95% CI 2-sided [0.84 to 1.07] — V116 Lot 1/V116 Lot 3
Statistical Analysis 39: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 19A: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.93, 95% CI 2-sided [0.82 to 1.04] — V116 Lot 2/V116 Lot 3
Statistical Analysis 40: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 20A: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.98, 95% CI 2-sided [0.84 to 1.14] — V116 Lot 1/V116 Lot 2
Statistical Analysis 41: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 20A: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.07, 95% CI 2-sided [0.92 to 1.24] — V116 Lot 1/V116 Lot 3
Statistical Analysis 42: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 20A: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.09, 95% CI 2-sided [0.94 to 1.27] — V116 Lot 2/V116 Lot 3
Statistical Analysis 43: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 22F: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.10, 95% CI 2-sided [0.93 to 1.29] — V116 Lot 1/V116 Lot 2
Statistical Analysis 44: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 22F: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.03, 95% CI 2-sided [0.87 to 1.21] — V116 Lot 1/V116 Lot 3
Statistical Analysis 45: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 22F: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.94, 95% CI 2-sided [0.80 to 1.10] — V116 Lot 2/V116 Lot 3
Statistical Analysis 46: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 23A: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cDLA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.85 to 1.17] — V116 Lot 1/V116 Lot 2
Statistical Analysis 47: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 23A: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.01, 95% CI 2-sided [0.86 to 1.19] — V116 Lot 1/V116 Lot 3
Statistical Analysis 48: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 23A: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.87 to 1.19] — V116 Lot 2/V116 Lot 3
Statistical Analysis 49: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 23B: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.22, 95% CI 2-sided [1.00 to 1.48] — V116 Lot 1/V116 Lot 2
Statistical Analysis 50: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 23B: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.98, 95% CI 2-sided [0.80 to 1.19] — V116 Lot 1/V116 Lot 3
Statistical Analysis 51: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 23B: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.80, 95% CI 2-sided [0.66 to 0.97] — V116 Lot 2/V116 Lot 3
Statistical Analysis 52: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 24F: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.88 to 1.18] — V116 Lot 1/V116 Lot 2
Statistical Analysis 53: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 24F: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.88 to 1.18] — V116 Lot 1/V116 Lot 3
Statistical Analysis 54: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 24F: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.01, 95% CI 2-sided [0.87 to 1.16] — V116 Lot 2/V116 Lot 3
Statistical Analysis 55: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 31: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.87 to 1.20] — V116 Lot 1/V116 Lot 2
Statistical Analysis 56: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 31: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.87 to 1.20] — V116 Lot 1/V116 Lot 3
Statistical Analysis 57: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 31: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.85 to 1.17] — V116 Lot 2/V116 Lot 3
Statistical Analysis 58: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 33F: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.11, 95% CI 2-sided [0.93 to 1.33] — V116 Lot 1/V116 Lot 2
Statistical Analysis 59: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 33F: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.08, 95% CI 2-sided [0.90 to 1.29] — V116 Lot 1/V116 Lot 3
Statistical Analysis 60: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 33F: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 0.97, 95% CI 2-sided [0.81 to 1.16] — V116 Lot 2/V116 Lot 3
Statistical Analysis 61: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 35B: GMT Ratio V116 Lot 1/V116 Lot 2; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.03, 95% CI 2-sided [0.91 to 1.17] — V116 Lot 1/V116 Lot 2
Statistical Analysis 62: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 35B: GMT Ratio V116 Lot 1/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.04, 95% CI 2-sided [0.91 to 1.18] — V116 Lot 1/V116 Lot 3
Statistical Analysis 63: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 35B: GMT Ratio V116 Lot 2/V116 Lot 3; Test type: Equivalence — Equivalence can be concluded if both the lower tailed and upper tailed p-values are < 0.025; p < 0.001, cLDA model — Identical p-values for the lower and upper bounds; [statistical method as in outcome 7, analysis 1]; GMT Ratio = 1.01, 95% CI 2-sided [0.89 to 1.14] — V116 Lot 2/V116 Lot 3

8. Secondary Outcome: GMTs of Serotype-specific OPA for All Serotypes in V116 Following Vaccination: Combined Lots of V116 or PPSV23
Description: Serotype-specific OPA titers for all serotypes in V116 following vaccination were determined using MOPA. Serotype-specific OPA GMTs and GMT ratios with 95% CI were calculated using a constrained longitudinal data analysis (cLDA) model. Per protocol, within-group CIs were not calculated.
Time Frame: Day 30
Population: All randomized participants without deviations from the protocol that may substantially affect the results of the immunogenicity endpoint and who had sufficient data to perform the analysis. Deviations include, but are not limited to the following: randomized but not vaccinated, blood drawn out of time window, prohibited concomitant medication or vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- V116 Combined Lots 1, 2 and 3: Participants received a single 0.5 mL IM dose of either V116 Lot 1, 2, or 3 on Day 1.
Arm/Group | V116 Combined Lots 1, 2 and 3 | PPSV23
Number analyzed (Participants) | 1617 | 540
Titers
  Serotype 3: number analyzed (Participants) | 1574 | 534
  Serotype 3 | 316.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 339.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 6A: number analyzed (Participants) | 1562 | 529
  Serotype 6A | 6491.7 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1866.4 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F: number analyzed (Participants) | 1580 | 531
  Serotype 7F | 6702.2 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5058.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 8: number analyzed (Participants) | 1585 | 537
  Serotype 8 | 3847.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4543.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9N: number analyzed (Participants) | 1590 | 533
  Serotype 9N | 18166.7 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 19031.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 10A: number analyzed (Participants) | 1586 | 534
  Serotype 10A | 7618.2 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5763.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 11A: number analyzed (Participants) | 1581 | 534
  Serotype 11A | 6494.4 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3728.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 12F: number analyzed (Participants) | 1583 | 534
  Serotype 12F | 7196.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5207.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15A: number analyzed (Participants) | 1520 | 512
  Serotype 15A | 10520.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2608.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15C: number analyzed (Participants) | 1571 | 529
  Serotype 15C | 11922.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4112.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 16F: number analyzed (Participants) | 1563 | 527
  Serotype 16F | 9415.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 2532.2 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 17F: number analyzed (Participants) | 1588 | 536
  Serotype 17F | 17330.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10159.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A: number analyzed (Participants) | 1593 | 533
  Serotype 19A | 3222.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3474.7 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 20A: number analyzed (Participants) | 1574 | 533
  Serotype 20A | 16183.8 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10994.2 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F: number analyzed (Participants) | 1573 | 530
  Serotype 22F | 11118.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8308.0 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23A: number analyzed (Participants) | 1550 | 519
  Serotype 23A | 8428.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1056.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23B: number analyzed (Participants) | 1583 | 533
  Serotype 23B | 2825.4 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 119.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 24F: number analyzed (Participants) | 1568 | 518
  Serotype 24F | 4892.9 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 250.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 31: number analyzed (Participants) | 1565 | 531
  Serotype 31 | 8865.6 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 654.5 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F: number analyzed (Participants) | 1576 | 533
  Serotype 33F | 35684.3 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 42515.6 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 35B: number analyzed (Participants) | 1578 | 537
  Serotype 35B | 12798.6 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3452.1 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 3: GMT Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMT Ratio = 0.93, 95% CI 2-sided [0.84 to 1.03] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 2: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 6A: GMT Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMT Ratio = 3.48, 95% CI 2-sided [3.01 to 4.02] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 3: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 7F: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 1.33, 95% CI 2-sided [1.18 to 1.49] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 4: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 8: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 0.85, 95% CI 2-sided [0.77 to 0.93] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 5: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 9N: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 0.95, 95% CI 2-sided [0.85 to 1.08] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 6: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 10A: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 1.32, 95% CI 2-sided [1.18 to 1.48] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 7: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 11A: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 1.74, 95% CI 2-sided [1.56 to 1.95] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 8: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 12F: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 1.38, 95% CI 2-sided [1.22 to 1.56] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 9: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 15A: GMT Ratio v116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 4.03, 95% CI 2-sided [3.56 to 4.56] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 10: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 15C: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 2.90, 95% CI 2-sided [2.49 to 3.38] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 11: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 16F: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 3.72, 95% CI 2-sided [3.32 to 4.17]; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 12: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 17F: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 1.71, 95% CI 2-sided [1.53 to 1.91] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 13: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 19A: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 0.93, 95% CI 2-sided [0.84 to 1.03] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 14: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 20A: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 1.47, 95% CI 2-sided [1.30 to 1.67] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 15: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 22F: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 1.34, 95% CI 2-sided [1.17 to 1.53] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 16: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 23A: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 7.98, 95% CI 2-sided [6.84 to 9.31] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 17: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 23B: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 23.72, 95% CI 2-sided [19.71 to 28.55] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 18: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 24F: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 19.55, 95% CI 2-sided [16.70 to 22.88] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 19: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 31: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 13.55, 95% CI 2-sided [11.68 to 15.71] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 20: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 33F: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 0.84, 95% CI 2-sided [0.73 to 0.97]; GMT Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 21: Comparison: V116 Combined Lots 1, 2 and 3 vs PPSV23; Serotype 35B: GMT Ratio V116 Combined Lots / PPSV23; Test type: Other; GMT Ratio = 3.71, 95% CI 2-sided [3.36 to 4.09] — V116 Combined Lots/PPSV23; GMT Ratio and 95% CI were estimated from a cLDA model

9. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Serotype-specific Immunoglobulin G (IgG) for All Serotypes in V116 Following Vaccination With Separate V116 Lots
Description: Serotype-specific IgG concentrations for all serotypes in V116 following vaccination were determined using pneumococcal electrochemiluminescence (PnECL). Serotype-specific pneumococcal IgG GMCs and GMC ratios with 95% confidence intervals were calculated using a cLDA model. Per protocol, within-group CIs were not calculated and the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Day 30
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 538 | 540 | 0
μg/mL
  Serotype 3: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 3 | 0.83 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.85 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.87 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 6A: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 6A | 5.94 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.84 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 7F: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 7F | 5.13 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 8: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 8 | 10.32 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10.52 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 10.42 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 9N: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 9N | 5.37 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.11 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.03 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 10A: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 10A | 9.63 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9.52 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 11A: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 11A | 6.33 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.28 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.21 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 12F: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 12F | 1.65 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.75 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.65 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 15A: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 15A | 13.63 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 13.00 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 14.20 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 15C: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 15C | 14.32 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 13.54 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 13.85 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 16F: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 16F | 1.77 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.96 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 17F: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 17F | 14.05 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 13.37 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 13.14 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 19A: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 19A | 7.70 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.94 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8.51 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 20A: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 20A | 13.54 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 14.18 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 14.09 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 22F: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 22F | 7.02 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.97 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 23A: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 23A | 4.26 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.34 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.34 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 23B: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 23B | 6.77 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.65 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.39 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 24F: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 24F | 4.32 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.55 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.34 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 31: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 31 | 3.47 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.94 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.47 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 33F: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 33F | 8.03 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.94 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 8.00 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
  Serotype 35B: number analyzed (Participants) | 532 | 535 | 536 | 0
  Serotype 35B | 11.84 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11.56 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 11.94 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. |
Statistical Analysis 1: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 3: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.98, 95% CI 2-sided [0.88 to 1.09] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 2: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 3: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.95, 95% CI 2-sided [0.85 to 1.05] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 3: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 3: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.97, 95% CI 2-sided [0.87 to 1.08] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 4: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 6A: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.12, 95% CI 2-sided [0.95 to 1.32] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 5: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 6A: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.02, 95% CI 2-sided [0.86 to 1.20] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 6: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 6A: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.91, 95% CI 2-sided [0.77 to 1.07] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 7: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 7F: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.97, 95% CI 2-sided [0.85 to 1.11] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 8: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 7F: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.03, 95% CI 2-sided [0.90 to 1.18] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 9: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 7F: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.06, 95% CI 2-sided [0.93 to 1.21] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 10: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 8: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.98, 95% CI 2-sided [0.86 to 1.12] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 11: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 8: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.87 to 1.13] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 12: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 8: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.89 to 1.15] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 13: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 9N: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.05, 95% CI 2-sided [0.91 to 1.21] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 14: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 9N: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.89, 95% CI 2-sided [0.77 to 1.03] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 15: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 9N: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.85, 95% CI 2-sided [0.74 to 0.98] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 16: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 10A: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.87 to 1.18] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 17: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 10A: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.97, 95% CI 2-sided [0.83 to 1.13] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 18: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 10A: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.95, 95% CI 2-sided [0.82 to 1.11] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 19: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 11A: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.90 to 1.14] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 20: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 11A: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.02, 95% CI 2-sided [0.91 to 1.15] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 21: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 11A: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.90 to 1.14] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 22: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 12F: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.95, 95% CI 2-sided [0.80 to 1.12] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 23: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 12F: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.00, 95% CI 2-sided [0.84 to 1.18] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 24: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 12F: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.06, 95% CI 2-sided [0.89 to 1.25] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 25: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 15A: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.05, 95% CI 2-sided [0.91 to 1.21] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 26: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 15A: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.96, 95% CI 2-sided [0.83 to 1.11] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 27: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 15A: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.92, 95% CI 2-sided [0.80 to 1.05] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 28: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 15C: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.06, 95% CI 2-sided [0.91 to 1.23] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 29: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 15C: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.03, 95% CI 2-sided [0.89 to 1.20] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 30: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 15C: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.98, 95% CI 2-sided [0.84 to 1.14] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 31: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 16F: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.90, 95% CI 2-sided [0.78 to 1.03] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 32: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 16F: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.90, 95% CI 2-sided [0.78 to 1.04] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 33: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 16F: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.88 to 1.15] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 34: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 17F: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.05, 95% CI 2-sided [0.91 to 1.21] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 35: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 17F: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.07, 95% CI 2-sided [0.93 to 1.23] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 36: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 17F: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.02, 95% CI 2-sided [0.88 to 1.17] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 37: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 19A: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.97, 95% CI 2-sided [0.85 to 1.11] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 38: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 19A: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.90, 95% CI 2-sided [0.79 to 1.04] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 39: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 19A: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.93, 95% CI 2-sided [0.82 to 1.07] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 40: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 20A: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.95, 95% CI 2-sided [0.83 to 1.10] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 41: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 20A: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.96, 95% CI 2-sided [0.84 to 1.10] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 42: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 20A: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.88 to 1.16] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 43: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 22F: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.87 to 1.16] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 44: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 22F: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.00, 95% CI 2-sided [0.87 to 1.16] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 45: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 22F: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.00, 95% CI 2-sided [0.86 to 1.15] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 46: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 23A: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.98, 95% CI 2-sided [0.84 to 1.16] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 47: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 23A: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.98, 95% CI 2-sided [0.83 to 1.15] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 48: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 23A: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.00, 95% CI 2-sided [0.85 to 1.17] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 49: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 23B: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.02, 95% CI 2-sided [0.87 to 1.18] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 50: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 23B: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.92, 95% CI 2-sided [0.79 to 1.07] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 51: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 23B: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.90, 95% CI 2-sided [0.77 to 1.05] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 52: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 24F: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.95, 95% CI 2-sided [0.80 to 1.13] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 53: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 24F: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.00, 95% CI 2-sided [0.84 to 1.19] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 54: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 24F: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.05, 95% CI 2-sided [0.88 to 1.25] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 55: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 31: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.77 to 1.00] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 56: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 31: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.00, 95% CI 2-sided [0.88 to 1.14] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 57: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 31: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 1.14, 95% CI 2-sided [1.00 to 1.30] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 58: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 33F: GMC Ratio V116 Lot 1/ V116 Lot 2; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.89 to 1.16] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 59: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 33F: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.00, 95% CI 2-sided [0.88 to 1.15] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 60: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 33F: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.87 to 1.13] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 61: Comparison: V116 Lot 1 vs V116 Lot 2; Serotype 35B: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 1.02, 95% CI 2-sided [0.90 to 1.17] — V116 Lot 1/V116 Lot 2; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 62: Comparison: V116 Lot 1 vs V116 Lot 3; Serotype 35B: GMC Ratio V116 Lot 1/ V116 Lot 3; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.87 to 1.13] — V116 Lot 1/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 63: Comparison: V116 Lot 2 vs V116 Lot 3; Serotype 35B: GMC Ratio V116 Lot 2/ V116 Lot 3; Test type: Other; GMC Ratio = 0.97, 95% CI 2-sided [0.85 to 1.10] — V116 Lot 2/V116 Lot 3; GMC Ratio and 95% CI were estimated from a cLDA model

10. Secondary Outcome: GMCs of Serotype-specific IgG for All Serotypes in V116 Following Vaccination: Combined Lots of V116 or PPSV23
Description: Serotype-specific IgG concentrations for all serotypes in V116 following vaccination were determined using PnECL. Serotype-specific pneumococcal IgG GMCs and GMC ratios with 95% confidence intervals were calculated using a cLDA model. Per protocol, within-group CIs were not calculated.
Time Frame: Day 30
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V116 Combined Lots 1, 2, and 3 | PPSV23
Number analyzed (Participants) | 1617 | 540
μg/mL
  Serotype 3: number analyzed (Participants) | 1603 | 539
  Serotype 3 | 0.85 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.77 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 6A: number analyzed (Participants) | 1603 | 539
  Serotype 6A | 5.67 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.45 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 7F: number analyzed (Participants) | 1603 | 539
  Serotype 7F | 5.19 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 3.36 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 8: number analyzed (Participants) | 1603 | 539
  Serotype 8 | 10.34 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 12.85 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 9N: number analyzed (Participants) | 1603 | 539
  Serotype 9N | 5.51 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.41 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 10A: number analyzed (Participants) | 1603 | 539
  Serotype 10A | 9.58 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 6.52 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 11A: number analyzed (Participants) | 1603 | 539
  Serotype 11A | 6.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.55 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 12F: number analyzed (Participants) | 1603 | 539
  Serotype 12F | 1.69 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.20 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15A: number analyzed (Participants) | 1603 | 539
  Serotype 15A | 13.55 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.99 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 15C: number analyzed (Participants) | 1603 | 539
  Serotype 15C | 13.90 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 4.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 16F: number analyzed (Participants) | 1603 | 539
  Serotype 16F | 1.91 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.30 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 17F: number analyzed (Participants) | 1603 | 539
  Serotype 17F | 13.46 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.28 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 19A: number analyzed (Participants) | 1603 | 539
  Serotype 19A | 8.01 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 7.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 20A: number analyzed (Participants) | 1603 | 539
  Serotype 20A | 13.82 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9.03 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 22F: number analyzed (Participants) | 1603 | 539
  Serotype 22F | 7.04 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 5.34 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23A: number analyzed (Participants) | 1603 | 539
  Serotype 23A | 4.29 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.53 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 23B: number analyzed (Participants) | 1603 | 539
  Serotype 23B | 6.96 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.21 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 24F: number analyzed (Participants) | 1603 | 539
  Serotype 24F | 4.44 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.31 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 31: number analyzed (Participants) | 1603 | 539
  Serotype 31 | 3.62 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 0.38 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 33F: number analyzed (Participants) | 1603 | 539
  Serotype 33F | 8.00 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 9.82 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
  Serotype 35B: number analyzed (Participants) | 1603 | 539
  Serotype 35B | 11.71 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated. | 1.66 [NA to NA] — NA means that per protocol, no within-group MOD were planned or calculated.
Statistical Analysis 1: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 3: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.10, 95% CI 2-sided [1.01 to 1.21] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 2: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 6A: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 3.91, 95% CI 2-sided [3.43 to 4.45] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 3: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 7F: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.54, 95% CI 2-sided [1.38 to 1.72] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 4: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 8: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 0.81, 95% CI 2-sided [0.73 to 0.89] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 5: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 9N: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.02, 95% CI 2-sided [0.91 to 1.14] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 6: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 10A: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.47, 95% CI 2-sided [1.30 to 1.66] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 7: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 11A: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.38, 95% CI 2-sided [1.26 to 1.52] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 8: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 12F: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.41, 95% CI 2-sided [1.23 to 1.62] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 9: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 15A: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 6.82, 95% CI 2-sided [6.08 to 7.65] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 10: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 15C: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 3.24, 95% CI 2-sided [2.86 to 3.67] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 11: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 16F: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 6.48, 95% CI 2-sided [5.83 to 7.19] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 12: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 17F: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.85, 95% CI 2-sided [1.66 to 2.07] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 13: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 19A: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.10, 95% CI 2-sided [0.98 to 1.22] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 14: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 20A: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.53, 95% CI 2-sided [1.37 to 1.71] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 15: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 22F: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 1.32, 95% CI 2-sided [1.17 to 1.49] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 16: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 23A: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 8.14, 95% CI 2-sided [7.19 to 9.23] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 17: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 23B: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 5.74, 95% CI 2-sided [5.08 to 6.48] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 18: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 24F: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 14.47, 95% CI 2-sided [12.77 to 16.40] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 19: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 31: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 9.55, 95% CI 2-sided [8.61 to 10.59] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 20: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 33F: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 0.81, 95% CI 2-sided [0.73 to 0.91] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model
Statistical Analysis 21: Comparison: V116 Combined Lots 1, 2, and 3 vs PPSV23; Serotype 35B: GMC Ratio V116 Combined Lots/ PPSV23; Test type: Other; GMC Ratio = 7.06, 95% CI 2-sided [6.41 to 7.77] — V116 Combined Lots/PPSV23; GMC Ratio and 95% CI were estimated from a cLDA model

11. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in Serotype-specific OPA for All Serotypes in V116 Following Vaccination With Separate V116 Lots
Description: Serotype-specific OPA GMFR for all serotypes in V116 following vaccination were determined using MOPA. The GMFR of each pneumococcal serotype was calculated as Day 30 GMT/Day 1 GMT. The 95% CIs were calculated based on based on the t-distribution. Per protocol, the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Baseline (Day 1) and Day 30
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 538 | 540 | 0
Ratio
  Serotype 3: number analyzed (Participants) | 413 | 427 | 429 | 0
  Serotype 3 | 8.2 [7.2 to 9.4] | 8.1 [7.2 to 9.1] | 8.2 [7.3 to 9.3] |
  Serotype 6A: number analyzed (Participants) | 366 | 393 | 403 | 0
  Serotype 6A | 46.8 [38.5 to 56.8] | 37.8 [31.1 to 45.9] | 35.8 [29.7 to 43.2] |
  Serotype 7F: number analyzed (Participants) | 438 | 435 | 428 | 0
  Serotype 7F | 17.6 [14.6 to 21.2] | 14.2 [11.8 to 17.0] | 14.8 [12.4 to 17.6] |
  Serotype 8: number analyzed (Participants) | 450 | 456 | 466 | 0
  Serotype 8 | 17.6 [14.7 to 21.1] | 16.2 [13.6 to 19.2] | 15.4 [12.9 to 18.5] |
  Serotype 9N: number analyzed (Participants) | 438 | 439 | 434 | 0
  Serotype 9N | 10.1 [8.8 to 11.7] | 10.4 [9.0 to 12.0] | 10.5 [9.0 to 12.2] |
  Serotype 10A: number analyzed (Participants) | 432 | 450 | 458 | 0
  Serotype 10A | 14.1 [11.8 to 16.7] | 15.2 [12.8 to 18.0] | 15.9 [13.3 to 18.9] |
  Serotype 11A: number analyzed (Participants) | 428 | 432 | 450 | 0
  Serotype 11A | 11.5 [9.5 to 14.0] | 11.3 [9.3 to 13.8] | 9.3 [7.8 to 11.1] |
  Serotype 12F: number analyzed (Participants) | 433 | 457 | 432 | 0
  Serotype 12F | 173.7 [144.8 to 208.5] | 152.0 [127.5 to 181.2] | 194.1 [162.5 to 231.7] |
  Serotype 15A: number analyzed (Participants) | 305 | 325 | 320 | 0
  Serotype 15A | 9.3 [7.8 to 11.2] | 8.8 [7.5 to 10.5] | 9.5 [7.9 to 11.3] |
  Serotype 15C: number analyzed (Participants) | 391 | 411 | 393 | 0
  Serotype 15C | 86.0 [68.7 to 107.8] | 78.8 [64.0 to 97.0] | 63.8 [51.2 to 79.5] |
  Serotype 16F: number analyzed (Participants) | 382 | 402 | 403 | 0
  Serotype 16F | 7.1 [6.2 to 8.2] | 7.6 [6.6 to 8.8] | 6.9 [6.2 to 7.8] |
  Serotype 17F: number analyzed (Participants) | 445 | 457 | 458 | 0
  Serotype 17F | 17.8 [15.3 to 20.9] | 18.5 [15.8 to 21.6] | 16.9 [14.4 to 19.8] |
  Serotype 19A: number analyzed (Participants) | 446 | 468 | 468 | 0
  Serotype 19A | 8.9 [7.7 to 10.3] | 8.5 [7.4 to 9.9] | 8.9 [7.8 to 10.3] |
  Serotype 20A: number analyzed (Participants) | 376 | 396 | 403 | 0
  Serotype 20A | 10.6 [9.1 to 12.3] | 11.7 [10.2 to 13.4] | 9.5 [8.3 to 10.8] |
  Serotype 22F: number analyzed (Participants) | 409 | 404 | 417 | 0
  Serotype 22F | 20.0 [16.1 to 24.7] | 15.4 [12.6 to 18.8] | 18.1 [14.9 to 22.0] |
  Serotype 23A: number analyzed (Participants) | 344 | 373 | 357 | 0
  Serotype 23A | 30.9 [24.8 to 38.4] | 27.7 [22.6 to 34.1] | 30.0 [24.5 to 36.7] |
  Serotype 23B: number analyzed (Participants) | 428 | 448 | 444 | 0
  Serotype 23B | 104.1 [85.2 to 127.2] | 91.0 [74.5 to 111.2] | 106.0 [87.2 to 128.8] |
  Serotype 24F: number analyzed (Participants) | 383 | 399 | 407 | 0
  Serotype 24F | 27.0 [22.2 to 32.9] | 24.0 [19.6 to 29.2] | 25.4 [20.8 to 31.0] |
  Serotype 31: number analyzed (Participants) | 383 | 406 | 398 | 0
  Serotype 31 | 25.1 [20.3 to 31.2] | 25.7 [20.9 to 31.6] | 21.2 [17.2 to 26.1] |
  Serotype 33F: number analyzed (Participants) | 393 | 411 | 425 | 0
  Serotype 33F | 13.1 [11.2 to 15.2] | 12.5 [10.7 to 14.5] | 12.3 [10.6 to 14.2] |
  Serotype 35B: number analyzed (Participants) | 420 | 434 | 441 | 0
  Serotype 35B | 4.6 [4.1 to 5.2] | 5.0 [4.4 to 5.7] | 4.7 [4.1 to 5.3] |

12. Secondary Outcome: Percentage of Participants With ≥4-fold Rise in Serotype-specific OPA for All Serotypes in V116 Following Vaccination With Separate V116 Lots
Description: Serotype-specific OPA titer were determined using MOPA. The percentage of participants with a ≥4-fold rise in serotype-specific OPA for all serotypes in V116 following vaccination were reported. The 95% CIs were calculated based on the exact binomial method proposed by Clopper and Pearson. Per protocol, the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Baseline (Day 1) and Day 30
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 538 | 540 | 0
Percentage of Participants
  Serotype 3: number analyzed (Participants) | 413 | 427 | 429 | 0
  Serotype 3 | 70.7 [66.1 to 75.1] | 71.0 [66.4 to 75.2] | 70.6 [66.1 to 74.9] |
  Serotype 6A: number analyzed (Participants) | 366 | 393 | 403 | 0
  Serotype 6A | 87.2 [83.3 to 90.4] | 86.5 [82.7 to 89.7] | 85.6 [81.8 to 88.9] |
  Serotype 7F: number analyzed (Participants) | 438 | 435 | 428 | 0
  Serotype 7F | 73.5 [69.1 to 77.6] | 69.7 [65.1 to 73.9] | 71.7 [67.2 to 75.9] |
  Serotype 8: number analyzed (Participants) | 450 | 456 | 466 | 0
  Serotype 8 | 72.7 [68.3 to 76.7] | 75.9 [71.7 to 79.7] | 70.4 [66.0 to 74.5] |
  Serotype 9N: number analyzed (Participants) | 438 | 439 | 434 | 0
  Serotype 9N | 69.6 [65.1 to 73.9] | 70.4 [65.9 to 74.6] | 72.1 [67.6 to 76.3] |
  Serotype 10A: number analyzed (Participants) | 432 | 450 | 458 | 0
  Serotype 10A | 70.6 [66.1 to 74.9] | 75.1 [70.8 to 79.0] | 73.8 [69.5 to 77.8] |
  Serotype 11A: number analyzed (Participants) | 428 | 432 | 450 | 0
  Serotype 11A | 64.3 [59.5 to 68.8] | 66.0 [61.3 to 70.4] | 61.3 [56.7 to 65.9] |
  Serotype 12F: number analyzed (Participants) | 433 | 457 | 432 | 0
  Serotype 12F | 94.5 [91.9 to 96.4] | 94.5 [92.0 to 96.4] | 95.6 [93.2 to 97.3] |
  Serotype 15A: number analyzed (Participants) | 305 | 325 | 320 | 0
  Serotype 15A | 66.9 [61.3 to 72.1] | 66.2 [60.7 to 71.3] | 67.5 [62.1 to 72.6] |
  Serotype 15C: number analyzed (Participants) | 391 | 411 | 393 | 0
  Serotype 15C | 87.5 [83.8 to 90.6] | 90.3 [87.0 to 93.0] | 88.3 [84.7 to 91.3] |
  Serotype 16F: number analyzed (Participants) | 382 | 402 | 403 | 0
  Serotype 16F | 66.0 [61.0 to 70.7] | 63.7 [58.8 to 68.4] | 62.5 [57.6 to 67.3] |
  Serotype 17F: number analyzed (Participants) | 445 | 457 | 458 | 0
  Serotype 17F | 82.0 [78.1 to 85.5] | 81.4 [77.5 to 84.9] | 80.8 [76.9 to 84.3] |
  Serotype 19A: number analyzed (Participants) | 446 | 468 | 468 | 0
  Serotype 19A | 65.2 [60.6 to 69.7] | 65.0 [60.4 to 69.3] | 66.2 [61.8 to 70.5] |
  Serotype 20A: number analyzed (Participants) | 376 | 396 | 403 | 0
  Serotype 20A | 72.3 [67.5 to 76.8] | 77.8 [73.4 to 81.8] | 72.7 [68.1 to 77.0] |
  Serotype 22F: number analyzed (Participants) | 409 | 404 | 417 | 0
  Serotype 22F | 76.3 [71.9 to 80.3] | 73.3 [68.7 to 77.5] | 78.4 [74.2 to 82.3] |
  Serotype 23A: number analyzed (Participants) | 344 | 373 | 357 | 0
  Serotype 23A | 79.7 [75.0 to 83.8] | 79.4 [74.9 to 83.4] | 82.1 [77.7 to 85.9] |
  Serotype 23B: number analyzed (Participants) | 428 | 448 | 444 | 0
  Serotype 23B | 91.4 [88.3 to 93.8] | 89.3 [86.0 to 92.0] | 90.3 [87.2 to 92.9] |
  Serotype 24F: number analyzed (Participants) | 383 | 399 | 407 | 0
  Serotype 24F | 78.9 [74.4 to 82.8] | 78.2 [73.8 to 82.2] | 76.7 [72.2 to 80.7] |
  Serotype 31: number analyzed (Participants) | 383 | 406 | 398 | 0
  Serotype 31 | 78.3 [73.9 to 82.4] | 79.1 [74.8 to 82.9] | 77.6 [73.2 to 81.6] |
  Serotype 33F: number analyzed (Participants) | 393 | 411 | 425 | 0
  Serotype 33F | 75.3 [70.7 to 79.5] | 73.2 [68.7 to 77.5] | 75.1 [70.7 to 79.1] |
  Serotype 35B: number analyzed (Participants) | 420 | 434 | 441 | 0
  Serotype 35B | 52.9 [48.0 to 57.7] | 49.5 [44.7 to 54.3] | 48.5 [43.8 to 53.3] |

13. Secondary Outcome: GMFR in Serotype-specific IgG for All Serotypes in V116 Following Vaccination With Separate V116 Lots
Description: Serotype-specific IgG GMFR for all serotypes in V116 following vaccination were determined using PnECL. The GMFR for each pneumococcal IgG serotype was calculated as Day 30 GMC/Day 1 GMC. The 95% CIs were calculated based on the t-distribution. Per protocol, the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Baseline (Day 1) and Day 30
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 538 | 540 | 0
Ratio
  Serotype 3: number analyzed (Participants) | 494 | 502 | 506 | 0
  Serotype 3 | 4.4 [4.0 to 4.8] | 4.7 [4.3 to 5.2] | 4.6 [4.1 to 5.0] |
  Serotype 6A: number analyzed (Participants) | 493 | 502 | 506 | 0
  Serotype 6A | 21.2 [18.7 to 24.1] | 18.8 [16.6 to 21.5] | 21.0 [18.7 to 23.7] |
  Serotype 7F: number analyzed (Participants) | 493 | 502 | 506 | 0
  Serotype 7F | 13.7 [12.3 to 15.2] | 13.4 [12.1 to 14.8] | 12.6 [11.3 to 14.0] |
  Serotype 8: number analyzed (Participants) | 493 | 502 | 506 | 0
  Serotype 8 | 14.3 [12.7 to 16.2] | 15.2 [13.5 to 17.0] | 14.5 [12.8 to 16.4] |
  Serotype 9N: number analyzed (Participants) | 493 | 502 | 505 | 0
  Serotype 9N | 15.9 [14.3 to 17.8] | 15.3 [13.6 to 17.3] | 17.1 [15.2 to 19.3] |
  Serotype 10A: number analyzed (Participants) | 494 | 501 | 506 | 0
  Serotype 10A | 15.0 [13.4 to 16.8] | 15.2 [13.5 to 17.1] | 15.7 [14.0 to 17.6] |
  Serotype 11A: number analyzed (Participants) | 494 | 502 | 506 | 0
  Serotype 11A | 7.2 [6.5 to 8.0] | 7.2 [6.5 to 8.0] | 7.0 [6.3 to 7.8] |
  Serotype 12F: number analyzed (Participants) | 494 | 502 | 505 | 0
  Serotype 12F | 16.3 [14.4 to 18.4] | 17.1 [15.1 to 19.3] | 15.8 [14.1 to 17.8] |
  Serotype 15A: number analyzed (Participants) | 492 | 502 | 505 | 0
  Serotype 15A | 23.1 [20.6 to 25.9] | 22.8 [20.4 to 25.5] | 23.4 [20.9 to 26.3] |
  Serotype 15C: number analyzed (Participants) | 494 | 502 | 505 | 0
  Serotype 15C | 28.5 [25.3 to 32.2] | 27.8 [24.7 to 31.3] | 27.3 [24.2 to 30.9] |
  Serotype 16F: number analyzed (Participants) | 493 | 502 | 505 | 0
  Serotype 16F | 8.4 [7.6 to 9.3] | 8.8 [7.9 to 9.9] | 9.1 [8.2 to 10.1] |
  Serotype 17F: number analyzed (Participants) | 494 | 502 | 506 | 0
  Serotype 17F | 23.5 [21.0 to 26.3] | 23.1 [20.6 to 25.9] | 21.5 [19.2 to 24.1] |
  Serotype 19A: number analyzed (Participants) | 494 | 502 | 506 | 0
  Serotype 19A | 5.5 [4.9 to 6.1] | 5.8 [5.2 to 6.4] | 6.0 [5.4 to 6.7] |
  Serotype 20A: number analyzed (Participants) | 494 | 502 | 504 | 0
  Serotype 20A | 9.2 [8.3 to 10.3] | 9.8 [8.8 to 10.9] | 9.8 [8.8 to 10.9] |
  Serotype 22F: number analyzed (Participants) | 493 | 502 | 506 | 0
  Serotype 22F | 20.4 [17.9 to 23.3] | 19.1 [16.6 to 22.0] | 19.4 [17.0 to 22.2] |
  Serotype 23A: number analyzed (Participants) | 492 | 502 | 504 | 0
  Serotype 23A | 20.3 [18.0 to 22.8] | 20.1 [17.9 to 22.5] | 20.3 [18.0 to 22.9] |
  Serotype 23B: number analyzed (Participants) | 492 | 502 | 505 | 0
  Serotype 23B | 13.9 [12.2 to 15.7] | 14.0 [12.2 to 16.0] | 15.0 [13.2 to 17.1] |
  Serotype 24F: number analyzed (Participants) | 492 | 502 | 506 | 0
  Serotype 24F | 14.7 [13.0 to 16.6] | 15.4 [13.6 to 17.5] | 14.6 [12.9 to 16.6] |
  Serotype 31: number analyzed (Participants) | 492 | 502 | 505 | 0
  Serotype 31 | 13.6 [12.3 to 15.0] | 15.7 [14.1 to 17.5] | 13.0 [11.7 to 14.5] |
  Serotype 33F: number analyzed (Participants) | 494 | 502 | 505 | 0
  Serotype 33F | 8.8 [7.9 to 9.8] | 9.1 [8.2 to 10.1] | 9.1 [8.2 to 10.0] |
  Serotype 35B: number analyzed (Participants) | 494 | 502 | 505 | 0
  Serotype 35B | 7.3 [6.5 to 8.1] | 7.3 [6.6 to 8.1] | 7.2 [6.5 to 8.0] |

14. Secondary Outcome: Percentage of Participants With ≥4-fold Rise in Serotype-specific IgG for All Serotypes in V116 Following Vaccination With Separate V116 Lots
Description: Serotype-specific IgG concentrations were determined using PnECL. The percentage of participants with a ≥4-fold rise in serotype-specific IgG for all serotypes in V116 were reported. The 95% CIs were calculated based on the exact binomial method proposed by Clopper and Pearson. Per protocol, the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Baseline (Day 1) and Day 30
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 538 | 540 | 0
Percentage of Participants
  Serotype 3: number analyzed (Participants) | 494 | 502 | 506 | 0
  Serotype 3 | 51.8 [47.3 to 56.3] | 54.4 [49.9 to 58.8] | 52.0 [47.5 to 56.4] |
  Serotype 6A: number analyzed (Participants) | 493 | 502 | 506 | 0
  Serotype 6A | 87.8 [84.6 to 90.6] | 85.3 [81.9 to 88.2] | 89.3 [86.3 to 91.9] |
  Serotype 7F: number analyzed (Participants) | 493 | 502 | 506 | 0
  Serotype 7F | 83.2 [79.6 to 86.4] | 84.1 [80.6 to 87.2] | 82.6 [79.0 to 85.8] |
  Serotype 8: number analyzed (Participants) | 493 | 502 | 506 | 0
  Serotype 8 | 80.5 [76.8 to 83.9] | 82.7 [79.1 to 85.9] | 81.4 [77.8 to 84.7] |
  Serotype 9N: number analyzed (Participants) | 493 | 502 | 505 | 0
  Serotype 9N | 86.0 [82.6 to 88.9] | 84.1 [80.6 to 87.2] | 82.8 [79.2 to 86.0] |
  Serotype 10A: number analyzed (Participants) | 494 | 501 | 506 | 0
  Serotype 10A | 82.8 [79.2 to 86.0] | 82.4 [78.8 to 85.7] | 83.4 [79.9 to 86.5] |
  Serotype 11A: number analyzed (Participants) | 494 | 502 | 506 | 0
  Serotype 11A | 67.4 [63.1 to 71.5] | 67.3 [63.0 to 71.4] | 63.8 [59.5 to 68.0] |
  Serotype 12F: number analyzed (Participants) | 494 | 502 | 505 | 0
  Serotype 12F | 83.8 [80.3 to 86.9] | 85.1 [81.6 to 88.1] | 84.4 [80.9 to 87.4] |
  Serotype 15A: number analyzed (Participants) | 492 | 502 | 505 | 0
  Serotype 15A | 91.1 [88.2 to 93.4] | 89.2 [86.2 to 91.8] | 90.3 [87.4 to 92.7] |
  Serotype 15C: number analyzed (Participants) | 494 | 502 | 505 | 0
  Serotype 15C | 90.9 [88.0 to 93.3] | 90.8 [88.0 to 93.2] | 90.1 [87.2 to 92.6] |
  Serotype 16F: number analyzed (Participants) | 493 | 502 | 505 | 0
  Serotype 16F | 73.2 [69.1 to 77.1] | 72.5 [68.4 to 76.4] | 74.7 [70.6 to 78.4] |
  Serotype 17F: number analyzed (Participants) | 494 | 502 | 506 | 0
  Serotype 17F | 90.3 [87.3 to 92.7] | 91.0 [88.2 to 93.4] | 87.7 [84.6 to 90.5] |
  Serotype 19A: number analyzed (Participants) | 494 | 502 | 506 | 0
  Serotype 19A | 58.5 [54.0 to 62.9] | 58.6 [54.1 to 62.9] | 59.3 [54.9 to 63.6] |
  Serotype 20A: number analyzed (Participants) | 494 | 502 | 504 | 0
  Serotype 20A | 72.9 [68.7 to 76.7] | 76.1 [72.1 to 79.8] | 74.8 [70.8 to 78.5] |
  Serotype 22F: number analyzed (Participants) | 493 | 502 | 506 | 0
  Serotype 22F | 84.2 [80.7 to 87.3] | 79.5 [75.7 to 82.9] | 84.2 [80.7 to 87.3] |
  Serotype 23A: number analyzed (Participants) | 492 | 502 | 504 | 0
  Serotype 23A | 89.0 [85.9 to 91.6] | 88.8 [85.8 to 91.5] | 86.3 [83.0 to 89.2] |
  Serotype 23B: number analyzed (Participants) | 492 | 502 | 505 | 0
  Serotype 23B | 77.6 [73.7 to 81.2] | 77.1 [73.2 to 80.7] | 78.6 [74.8 to 82.1] |
  Serotype 24F: number analyzed (Participants) | 492 | 502 | 506 | 0
  Serotype 24F | 81.1 [77.4 to 84.5] | 80.9 [77.2 to 84.2] | 79.6 [75.9 to 83.1] |
  Serotype 31: number analyzed (Participants) | 492 | 502 | 505 | 0
  Serotype 31 | 85.8 [82.4 to 88.7] | 84.3 [80.8 to 87.3] | 82.4 [78.8 to 85.6] |
  Serotype 33F: number analyzed (Participants) | 494 | 502 | 505 | 0
  Serotype 33F | 73.5 [69.4 to 77.3] | 71.7 [67.6 to 75.6] | 73.7 [69.6 to 77.5] |
  Serotype 35B: number analyzed (Participants) | 494 | 502 | 505 | 0
  Serotype 35B | 67.8 [63.5 to 71.9] | 66.7 [62.4 to 70.8] | 64.2 [59.8 to 68.3] |

15. Secondary Outcome: GMTs of Serotype-specific OPA for Cross-reactive Serotypes Following Vaccination With Separate V116 Lots
Description: Serotype-specific OPA titers for cross-reactive serotypes (6A, 6C, 15B, and 15C) were determined using MOPA. The 95% CIs for serotype-specific OPA GMTs were calculated based on based on the t-distribution. Per protocol, the PPSV23 treatment group was not included as it was not analyzed with the individual lots of V116.
Time Frame: Day 30
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
Number analyzed (Participants) | 539 | 538 | 540 | 0
Titers
  Serotype 6A: number analyzed (Participants) | 428 | 451 | 442 | 0
  Serotype 6A | 6849.6 [6120.8 to 7665.0] | 6009.2 [5348.8 to 6751.0] | 6724.3 [5967.6 to 7577.0] |
  Serotype 6C: number analyzed (Participants) | 434 | 442 | 438 | 0
  Serotype 6C | 3972.7 [3501.8 to 4506.9] | 3421.5 [3006.5 to 3893.8] | 3750.9 [3298.0 to 4265.9] |
  Serotype 15B: number analyzed (Participants) | 416 | 437 | 417 | 0
  Serotype 15B | 11799.5 [10317.9 to 13493.8] | 10062.4 [8838.3 to 11456.1] | 11139.5 [9619.7 to 12899.4] |
  Serotype 15C: number analyzed (Participants) | 429 | 442 | 422 | 0
  Serotype 15C | 13079.8 [11543.5 to 14820.6] | 11332.5 [9905.9 to 12964.7] | 11290.9 [9805.6 to 13001.2] |

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected up to 30 days postvaccination. Serious adverse events and all-cause mortality were reported throughout the duration of the study, up to 194 days.
Description: The analysis population for All-Cause Mortality included all randomized participants. The safety analysis population included all randomized participants who received the study vaccination according to the vaccination they received. One participant randomized to the V116 Lot 1 arm incorrectly received V116 Lot 3, one participant randomized into the V116 Lot 2 arm incorrectly received V116 Lot 1,and one participant randomized into the V116 Lot 2 arm incorrectly received PPSV23.
Arm/Group | V116 Lot 1 | V116 Lot 2 | V116 Lot 3 | PPSV23
All-Cause Mortality (participants affected / at risk) | 0/541 | 0/540 | 0/541 | 1/540
Serious Adverse Events (participants affected / at risk) | 8/539 | 5/536 | 1/541 | 6/541
Other Adverse Events (participants affected / at risk) | 428/539 | 415/536 | 421/541 | 388/541
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 Lot 1 (N=539) | V116 Lot 2 (N=536) | V116 Lot 3 (N=541) | PPSV23 (N=541)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 Lot 1 (N=539) | V116 Lot 2 (N=536) | V116 Lot 3 (N=541) | PPSV23 (N=541)
Fatigue (General disorders) | 206 (206) | 184 (186) | 187 (188) | 184 (186)
Injection site erythema (General disorders) | 74 (74) | 79 (80) | 71 (71) | 41 (41)
Injection site pain (General disorders) | 393 (394) | 391 (392) | 400 (401) | 328 (328)
Injection site swelling (General disorders) | 68 (68) | 82 (82) | 64 (64) | 41 (41)
Myalgia (Musculoskeletal and connective tissue disorders) | 98 (98) | 75 (75) | 95 (95) | 49 (49)
Headache (Nervous system disorders) | 165 (172) | 154 (166) | 154 (163) | 131 (140)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. In this case, a coordinating investigator will be designated by mutual agreement. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT05464420/Prot_SAP_000.pdf